CLINICAL TRIAL: NCT00281918
Title: Phase III Trial of Combined Immunochemotherapy With Fludarabine, Cyclophosphamide and Rituximab (FCR) Versus Chemotherapy With Fludarabine and Cyclophosphamide (FC) Alone in Patients With Previously Untreated Chronic Lymphocytic Leukaemia
Brief Title: Fludarabine and Cyclophosphamide With or Without Rituximab in Patients With Previously Untreated Chronic B-Cell Lymphocytic Leukemia
Acronym: CLL-8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: German CLL Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454560; GCLLSG-CLL-8; EU-20560; ML17102
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Results first posted 2011-03-29 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Leukemia
Keywords: B-cell chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Cyclophosphamide; fludarabine phosphate

ARMS (2):
- Fludarabine+Cyclophosphamide+Rituximab (FCR) (Experimental)
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate
- Fludarabine+Cyclophosphamide (FC) (Active Comparator)
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine Phosphate

INTERVENTIONS:
Drug: Rituximab — Intravenous repeating dose
  Arms: Fludarabine+Cyclophosphamide+Rituximab (FCR)
Drug: Cyclophosphamide — Intravenous repeating dose
Drug: Fludarabine Phosphate — Intravenous repeating dose

SUMMARY:
This randomized phase III trial is studying fludarabine, cyclophosphamide, and rituximab to see how well they work compared to fludarabine and cyclophosphamide in treating patients with B-cell chronic lymphocytic leukemia.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed B-cell chronic lymphocytic leukemia (CLL) defined by the National Cancer Institute (NCI) Working Group criteria
* Meets 1 of the following criteria:

  * Binet stage C disease
  * Binet stage B disease AND ≥ 1 of the following signs or symptoms*:

    * B symptoms (night sweats, weight loss ≥ 10% within the previous 6 months, fevers > 38°C or 100.4°F for ≥ 2 weeks without evidence of infection), or constitutional symptoms (fatigue)
    * Continuous progression (doubling of peripheral lymphocyte count within the past 6 months and absolute lymphocyte count > 50 G/I)
    * Evidence of progressive marrow failure as manifested by the development/worsening of anemia and/or thrombocytopenia
    * Massive, progressive or painful splenomegaly or hypersplenism
    * Massive lymph nodes or lymph node clusters (> 10 cm in longest diameter), danger of organ complications through large lymphoma (e.g., vascular compression or tracheal narrowing), or progressive lymphadenopathy
    * Occurrence of symptomatic hyperviscosity problems at leukocyte counts > 200 G/I (symptomatic leukostasis) NOTE: * Marked hypogammaglobulinemia or the development of a monoclonal protein in the absence of any of the above criteria for active disease is not sufficient for eligibility
* No Binet stage A disease
* No transformation to an aggressive B-cell malignancy (e.g., diffuse large cell lymphoma, Richter's syndrome, or prolymphocytic leukemia)

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Cumulative Illness Rating Scale (CIRS) score > 6
* Life expectancy > 6 months
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* Alkaline phosphatase and transaminases ≤ 2 times ULN
* Creatinine clearance ≥ 70 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study treatment
* No known hypersensitivity with anaphylactic reaction to humanized monoclonal antibodies or any of the study drugs
* No cerebral dysfunction that precludes chemotherapy
* No active bacterial, viral, or fungal infection
* No clinically significant autoimmune cytopenia or Coombs-positive hemolytic anemia
* No other active malignancy requiring concurrent treatment except basal cell carcinoma or tumors treated curatively by surgery
* No medical or psychological condition that would preclude study therapy
* No concurrent disease that requires prolonged (> 1 month) therapy involving glucocorticoids

PRIOR CONCURRENT THERAPY:

* No previous treatment of CLL by chemotherapy, radiotherapy, or immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 817 (Actual)
Dates: Start 2003-07; Primary Completion 2007-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hallek, MD, Study Chair — Medizinische Universitaetsklinik I at the University of Cologne
Locations (162):
- Australia (6):
  - Gosford Hospital, Gosford, New South Wales
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead - Wentworthville, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Frankston Hospital, Frankston, Victoria
- Austria (3):
  - Allg. Krankenhaus der Stadt Wien Universitaets-Kinderklinik, Vienna
  - Hanuschkrankenhaus, Vienna
  - Rudolfinerhaus, Vienna
- Belgium (6):
  - AZ Sint-Jan, Bruges
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
  - Clinique Universitaire De Mont-Godinne, Mont-Godinne Yvoir
- Czechia (5):
  - Masaryk University Hospital, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - University Hospital - Olomouc, Olomouc
  - University Hospital in Pilsen - Lochotin, Pilsen-Lochotin
  - First Medical Clinic of Charles University Hospital, Prague
- Denmark (2):
  - Copenhagen County Herlev University Hospital, Copenhagen
  - Vejle Sygehus, Vejle
- France (6):
  - Hopital Louis Pasteur, Colmar
  - Hopital Andre Mignot, Le Chesnay
  - Centre Leon Berard, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez
- Germany (118):
  - Praxis Fur Hamatologie und Onkologie Ahaus, Ahaus
  - Gemeinschaftspraxis Fuer Innere Medizin, Haematologie Und Internistische Onkologie, Ansbach
  - Hamatologische/Onkologische Gemeinschaftspraxis - Augsburg, Augsburg
  - Klinikum Augsburg, Augsburg
  - Humaine - Clinic, Bad Saarow
  - Internistische Praxis - Bayreuth, Bayreuth
  - Internistische Gemeinschaftspraxis - Berlin, Berlin
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld
  - Krankenhaus Bietigheim, Bietigheim
  - Augusta-Kranken-Anstalt gGmbH, Bochum
  - Marienhospital Bottrop gGmbH, Bottrop
  - DIAKO Ev. Diakonie Krankenhaus gGmbH, Bremen
  - Krankenhaus Burglengenfeld, Burglengenfeld
  - Onkologische Schwerpunktpraxis at Facharzt fuer Innere Medizin, Coesfeld
  - Praxis Fuer Haematologie Internistische Onkologie, Cologne
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Onkologische Schwerpunktpraxis, Cottbus
  - Onkologische Gemeinschaftspraxis - Dresden, Dresden
  - Internistische Praxis - Dusseldorf, Düsseldorf
  - Florence-Nightingale-Krankenhause, Deaconess Kaiserswerth, Düsseldorf
  - Krankenhaus Benrath, Düsseldorf
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - St. Georg Klinikum Eisenach GmbH, Eisenach
  - Helios Klinikum Erfurt, Erfurt
  - Internistiche Praxis, Erfurt
  - Onkologische Schwerpunkt Praxis, Erlangen
  - St. Antonius Hospital, Eschweiler
  - Universitaetsklinikum Essen, Essen
  - Evangelisches Krankenhaus Essen Werden, Essen
  - Staedtische Kliniken Esslingen, Esslingen am Neckar
  - Internistische Gemeinschaftspraxis - Forchheim, Forchheim
  - Staedtische Kliniken Frankfurt am Main - Hoechst, Frankfurt
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Gemeinschaftspraxis - Freiburg, Freiburg im Breisgau
  - Klinikum Garmisch - Partenkirchen GmbH, Garmisch-Partenkirchen
  - Internistische Praxis - Gerlingen, Gerlingen
  - Gemeinschaftspraxis Fuer Innere Medizin, Hematologie Und Onkologie, Giessen
  - Universitaetsklinikum Goettingen, Göttingen
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - St. Marien Hospital - Katholisches Krankenhaus Hagen gGmbH, Hagen
  - Internistische Praxis - Halle, Halle
  - Universitaetsklinikum Halle, Halle
  - Asklepios Klinik St. Georg, Hamburg
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - St. Marien-Hospital Hamm - Klinik Knappenstrasse, Hamm
  - Evangelische Krankenhaus Hamm, Hamm
  - Krankenhaus Siloah - Medizinische Klinik II, Hanover
  - Universitatsklinikum Heidelberg, Heidelberg
  - Marienhospital at Ruhr University Bochum, Herne
  - Privatklinik Dr. R. Schindlbeck GmbH & Co. KG, Herrsching am Ammersee
  - Universitaetsklinikum des Saarlandes, Homburg
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - Gemeinschaftspraxis Innere Medizin, Jena
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - St. Vincentius-Kliniken, Karlsruhe
  - Internistische Gemeinschaftspraxis - Kassel, Kassel
  - Klinikum Kempten Oberallgaeu, Kempten
  - Internistische Praxis - Kiel, Kiel
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Praxis fuer Haematologie und Onkologie, Koblenz
  - Stiftungsklinikum Mittelrhein - Gesundheitszentrum Evangelisches Stift Sankt Martin Koblenz gGmbH, Koblez
  - Internistische Onkologische Praxis - Kronach, Kronach
  - Klinikum Landshut, Landshut
  - Onkologische Schwerpunktpraxis - Leer, Leer
  - Klinikum "St. Georg" Leipzig, Leipzig
  - Klinikum Lippe - Lemgo, Lemgo
  - Internistische Praxis - Loerrach, Loerrach
  - Gemeinschaftspraxis - Ludwigshafen, Ludwigshafen
  - Sana Kliniken Luebeck, Lübeck
  - Internistische Gemeinschaftspraxis - Magdeburg, Magdeburg
  - Staedtisches Klinikum Magdeburg - Altstadt, Magdeburg
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - Universitatsklinik Mainz, Mainz
  - III Medizinische Klinik Mannheim, Mannheim
  - Krankenhaus Maria Hilf GmbH, Mönchengladbach
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Staedtisches Krankenhaus Muenchen - Harlaching, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Haematologische Schwerpunktpraxis, Munich
  - Hamatologie/Onkologie Praxisgemeinschaft - Muenchen, München
  - University of Muenster, Münster
  - Haematologisch - Onkologische Gemeinschaftspraxis, Münster
  - Onkologische Schwerpunktpraxis Dr. Schmidt, Neunkirchen
  - Praxis fuer Haematologie und Interne Onkologie, Norderstedt
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
  - Gemeinschaftspraxis - Oberhausen, Oberhausen
  - Internistische Gemeinschaftspraxis - Offenbach, Offenbach
  - Internistische Gemeinschaftspraxis - Oldenburg, Oldenburg
  - Klinikum Oldenburg, Oldenburg
  - Asklepios Klinik Pasewalk, Pasewalk
  - Municipal Hospital Complex, Pforzheim
  - Klinikum Ernst Von Bergmann, Potsdam
  - Elisabeth Krankenhaus, Recklinghausen
  - Krankenhaus Barmherzige Brueder Regensburg, Regensburg
  - Klinik und Poliklinik fuer Innere Medizin - Universitaet Rostock, Rostock
  - Caritasklinik St. Theresia, Saarbrücken
  - Nordwestkrankenhaus Sanderbusch, Sanderbusch
  - St. Marien - Krankenhaus Siegen GMBH, Siegen
  - Internistische Gemeinschaftspraxis - Stuttgart, Stuttgart
  - Haematologische Praxis, Stuttgart
  - Klinik fuer Onkologie - Katharinenhospital Stuttgart, Stuttgart
  - Diakonie Klinikum Stuttgart, Stuttgart
  - Marienhospital Stuttgart, Stuttgart
  - KKH Torgau, Torgau
  - Onkologische Gemeinschaftspraxis - Trier, Trier
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Praxis Fuer Internistische Haematologie / Onkologie, Troisdorf
  - Universitaetsklinikum Tuebingen, Tübingen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - Municipal Hospital Complex, Villingen-Schwenningen
  - Praxis fur Innere Medizin - Wanzleben, Wanzleben
  - Haematologische Praxis, Weiden
  - Schwerpunktpraxis Hamatologie/Onkologie - Wesel, Wesel
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
  - Kliniken St. Antonius, Wuppertal
  - Hamatologisch - Onkologische Praxis Wurzburg, Würzburg
  - Medizinische Klinik und Poliklinik II - Universitaetsklinikum Wuerzburg, Würzburg
- Israel (6):
  - Soroka University Medical Center, Beersheba
  - BNAI Zion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Hadassah University Hospital, Jerusalem
  - Riverview Cancer Care Medical Associates, PC, Kfar Saba
  - Kaplan Hospital, Rehovot
- Italy (5):
  - Ospedale Oncologico A. Businco, Cagliari
  - Fondazione Centro San Raffaele Del Monte Tabor, Milan
  - Perugia Regional Cancer Center, Perugia
  - Ospedale Sant' Eugenio, Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Canterbury Health Laboratories, Christchurch
  - Palmerston North Hospital, Palmerston North
- Spain (2):
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Virgen Del La Salud, Toledo

REFERENCES:
- [Derived] Langerbeins P, Giza A, Robrecht S, Cramer P, von Tresckow J, Al-Sawaf O, Fink AM, Furstenau M, Kutsch N, Simon F, Goede V, Hoechstetter M, Niemann CU, da Cunha-Bang C, Kater A, Dubois J, Gregor M, Staber PB, Tausch E, Schneider C, Stilgenbauer S, Eichhorst B, Fischer K, Hallek M. Reassessing the chronic lymphocytic leukemia International Prognostic Index in the era of targeted therapies. Blood. 2024 Jun 20;143(25):2588-2598. doi: 10.1182/blood.2023022564. PMID 38620092
- [Derived] Bloehdorn J, Krzykalla J, Holzmann K, Gerhardinger A, Jebaraj BMC, Bahlo J, Humphrey K, Tausch E, Robrecht S, Mertens D, Schneider C, Fischer K, Hallek M, Dohner H, Benner A, Stilgenbauer S. Integrative prognostic models predict long-term survival after immunochemotherapy in chronic lymphocytic leukemia patients. Haematologica. 2022 Mar 1;107(3):615-624. doi: 10.3324/haematol.2020.251561. PMID 33730841
- [Derived] Jaramillo S, Agathangelidis A, Schneider C, Bahlo J, Robrecht S, Tausch E, Bloehdorn J, Hoechstetter M, Fischer K, Eichhorst B, Goede V, Hallek M, Dohner H, Rosenquist R, Ghia P, Stamatopoulos K, Stilgenbauer S. Prognostic impact of prevalent chronic lymphocytic leukemia stereotyped subsets: analysis within prospective clinical trials of the German CLL Study Group (GCLLSG). Haematologica. 2020 Nov 1;105(11):2598-2607. doi: 10.3324/haematol.2019.231027. PMID 33131249
- [Derived] Kreuzberger N, Damen JA, Trivella M, Estcourt LJ, Aldin A, Umlauff L, Vazquez-Montes MD, Wolff R, Moons KG, Monsef I, Foroutan F, Kreuzer KA, Skoetz N. Prognostic models for newly-diagnosed chronic lymphocytic leukaemia in adults: a systematic review and meta-analysis. Cochrane Database Syst Rev. 2020 Jul 31;7(7):CD012022. doi: 10.1002/14651858.CD012022.pub2. PMID 32735048
- [Derived] Dimier N, Delmar P, Ward C, Morariu-Zamfir R, Fingerle-Rowson G, Bahlo J, Fischer K, Eichhorst B, Goede V, van Dongen JJM, Ritgen M, Bottcher S, Langerak AW, Kneba M, Hallek M. A model for predicting effect of treatment on progression-free survival using MRD as a surrogate end point in CLL. Blood. 2018 Mar 1;131(9):955-962. doi: 10.1182/blood-2017-06-792333. Epub 2017 Dec 18. PMID 29255066
- [Derived] Fischer K, Bahlo J, Fink AM, Goede V, Herling CD, Cramer P, Langerbeins P, von Tresckow J, Engelke A, Maurer C, Kovacs G, Herling M, Tausch E, Kreuzer KA, Eichhorst B, Bottcher S, Seymour JF, Ghia P, Marlton P, Kneba M, Wendtner CM, Dohner H, Stilgenbauer S, Hallek M. Long-term remissions after FCR chemoimmunotherapy in previously untreated patients with CLL: updated results of the CLL8 trial. Blood. 2016 Jan 14;127(2):208-15. doi: 10.1182/blood-2015-06-651125. Epub 2015 Oct 20. PMID 26486789
- [Derived] Weisser M, Yeh RF, Duchateau-Nguyen G, Palermo G, Nguyen TQ, Shi X, Stinson SY, Yu N, Dufour A, Robak T, Salogub GN, Dmoszynska A, Solal-Celigny P, Warzocha K, Loscertales J, Catalano J, Larratt L, Rossiev VA, Bence-Bruckler I, Geisler CH, Montillo M, Fischer K, Fink AM, Hallek M, Bloehdorn J, Busch R, Benner A, Dohner H, Valente N, Wenger MK, Stilgenbauer S, Dornan D. PTK2 expression and immunochemotherapy outcome in chronic lymphocytic leukemia. Blood. 2014 Jul 17;124(3):420-5. doi: 10.1182/blood-2013-12-538975. Epub 2014 Jun 10. PMID 24916506
- [Derived] Pflug N, Bahlo J, Shanafelt TD, Eichhorst BF, Bergmann MA, Elter T, Bauer K, Malchau G, Rabe KG, Stilgenbauer S, Dohner H, Jager U, Eckart MJ, Hopfinger G, Busch R, Fink AM, Wendtner CM, Fischer K, Kay NE, Hallek M. Development of a comprehensive prognostic index for patients with chronic lymphocytic leukemia. Blood. 2014 Jul 3;124(1):49-62. doi: 10.1182/blood-2014-02-556399. Epub 2014 May 5. PMID 24797299
- [Derived] Stilgenbauer S, Schnaiter A, Paschka P, Zenz T, Rossi M, Dohner K, Buhler A, Bottcher S, Ritgen M, Kneba M, Winkler D, Tausch E, Hoth P, Edelmann J, Mertens D, Bullinger L, Bergmann M, Kless S, Mack S, Jager U, Patten N, Wu L, Wenger MK, Fingerle-Rowson G, Lichter P, Cazzola M, Wendtner CM, Fink AM, Fischer K, Busch R, Hallek M, Dohner H. Gene mutations and treatment outcome in chronic lymphocytic leukemia: results from the CLL8 trial. Blood. 2014 May 22;123(21):3247-54. doi: 10.1182/blood-2014-01-546150. Epub 2014 Mar 20. PMID 24652989
- [Derived] Eichhorst BF, Fischer K, Fink AM, Elter T, Wendtner CM, Goede V, Bergmann M, Stilgenbauer S, Hopfinger G, Ritgen M, Bahlo J, Busch R, Hallek M; German CLL Study Group (GCLLSG). Limited clinical relevance of imaging techniques in the follow-up of patients with advanced chronic lymphocytic leukemia: results of a meta-analysis. Blood. 2011 Feb 10;117(6):1817-21. doi: 10.1182/blood-2010-04-282228. Epub 2010 Dec 7. PMID 21139079
- [Derived] Hallek M, Fischer K, Fingerle-Rowson G, Fink AM, Busch R, Mayer J, Hensel M, Hopfinger G, Hess G, von Grunhagen U, Bergmann M, Catalano J, Zinzani PL, Caligaris-Cappio F, Seymour JF, Berrebi A, Jager U, Cazin B, Trneny M, Westermann A, Wendtner CM, Eichhorst BF, Staib P, Buhler A, Winkler D, Zenz T, Bottcher S, Ritgen M, Mendila M, Kneba M, Dohner H, Stilgenbauer S; International Group of Investigators; German Chronic Lymphocytic Leukaemia Study Group. Addition of rituximab to fludarabine and cyclophosphamide in patients with chronic lymphocytic leukaemia: a randomised, open-label, phase 3 trial. Lancet. 2010 Oct 2;376(9747):1164-74. doi: 10.1016/S0140-6736(10)61381-5. PMID 20888994

RESULTS

PARTICIPANT FLOW:
Groups:
- Fludarabine+Cyclophosphamide (FC): Fludarabine+cyclophosphamide (FC) intravenously for a total of 6 treatment cycles at intervals of 28 days. Fludarabine: 25 mg/m² IV on Days 1, 2, 3 for 6 cycles. Cyclophosphamide: 250 mg/m² IV on Days 1, 2, 3 for 6 cycles.
- Fludarabine+Cyclophosphamide+Rituximab (FCR): Rituximab intravenously for a total of 6 treatment cycles at intervals of 28 days. Cycle 1: 375 mg/m² IV on Day 0; Cycles 2-6: 500 mg/m² IV on Day 1. FC intravenously for a total of 6 treatment cycles at intervals of 28 days. Fludarabine: 25 mg/m² IV over 15-30 min on Days 1, 2, 3 for 6 cycles. Cyclophosphamide: 250 mg/m² IV over 15-30 min on Days 1, 2, 3 for 6 cycles.
Period: Overall Study
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Started | 409 (Informed consent unavailable for 2 patients at time of analysis; intent-to-treat population was 407.) | 408 (Informed consent unavailable for 5 patients at time of analysis; intent-to-treat population was 403.)
Safety Population; Received Study Drug | 398 | 402
Completed | 267 (Completed all 6 cycles of study medication.) | 300 (Completed all 6 cycles of study medication.)
Not Completed | 142 | 108

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR) | Total
Number analyzed (Participants) | 407 | 403 | 810
Age Continuous [Mean (Standard Deviation); unit: years] | 59.3 (8.55) | 59.6 (8.70) | 59.5 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 105 | 210
  Male | 302 | 298 | 600

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time between randomization and the date of first documented disease progression, relapse or death by any cause, whichever came first.
Time Frame: Median observation time at time of analysis was approximately 21 months
Population: The Intent-to-treat (ITT) population was comprised of all patients randomized in the study, irrespective of whether they received treatment or not. Informed consent was unavailable at the time of analysis for 2 patients in the FC group and 5 patients in the FCR group. ITT population: FC = 407; FCR = 403.
Measure: Median (Full Range); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 407 | 403
Days | 981.0 [1 to 1343] | 1212.0 [1 to 1372]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p < .0001, Log Rank

2. Secondary Outcome: Event-free Survival (EFS)
Description: Event-free survival (EFS) was defined as the time between randomization and the date of disease progression, relapse, start of new CLL treatment or death by any cause.
Time Frame: Median observation time at time of analysis was approximately 21 months
Population: The ITT population was comprised of all patients randomized in the study, irrespective of whether they received treatment or not. Informed consent was unavailable at the time of analysis for 2 patients in the FC group and 5 patients in the FCR group. ITT population: FC = 407; FCR = 403.
Measure: Median (Full Range); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 407 | 403
Days | 947.0 [1 to 1343] | 1212.0 [1 to 1372]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p < .0001, Log Rank

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time between randomization and the date of death due to any cause. Median OS was not reached.
Time Frame: Median observation time at time of analysis was approximately 21 months
Population: as for outcome 2
Measure: Number; unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 407 | 403
Days
  Minimum number of days to an event | 5 [83 to 90] | 4 [89 to 95]
  Maximum number of days to an event | 1373 | 1372
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p = 0.0427, Log Rank

4. Secondary Outcome: Disease-free Survival (DFS) of Patients With Confirmed Complete Response (CR).
Description: CR is defined by at least 8 weeks of: 1)Absence of lymphadenopathy 2)No hepatomegaly or splenomegaly 3)Absence of B-symptoms 4)Normal blood count 5)Bone marrow aspirate and biopsy 8 weeks after the clinical and laboratory results demonstrated that a CR was achieved. A marrow sample had to be normocellular for age with less than 30% lymphocytes. Lymphoid nodules had to be absent. If marrow was hypocellular,a repeat biopsy was taken 4 weeks later and samples were re-reviewed in conjunction with the prior pathology. DFS was calculated from time of CR to relapse or death. Median DFS was not reached.
Time Frame: Median observation time at time of analysis was approximately 21 months
Population: as for outcome 2
Measure: Number; unit: Days to an event
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 407 | 403
Days to an event
  Minimum number of days to an event | 84 [0 to 0] | 91 [939 to 9999]
  Maximum number of days to an event | 1164 | 1226
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p = 0.7882, Log Rank

5. Primary Outcome: Final Analysis: Time to Progression-free Survival Event
Description: Progression-free survival was defined as the time between randomization and the date of first documented disease progression, relapse or death by any cause, whichever came first.
Time Frame: Median observation time was approximately 66.4 months
Population: Participants from the Intent-to-treat population, that included all randomized participants, with PFS events.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 297 | 253
Days | 998.0 [886 to 1129] | 1703.0 [1543 to 1853]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p < .0001, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.48 to 0.67]

6. Secondary Outcome: Final Analysis: Time to Overall Survival Event
Description: Overall survival (OS) was defined as the time between randomization and the date of death due to any cause.
Time Frame: Median observation time was approximately 66.4 months
Population: Participants from the Intent-to-treat population, that included all randomized participants who died.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 154 | 125
Days | 2613.0 [2354 to NA] — Upper limit of the 95% confidence interval has not been reached. | NA [2745 to NA] — Median time to event and upper limit of the 95% confidence have not been reached.
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p = 0.0010, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.54 to 0.86]

7. Secondary Outcome: Final Analysis: Time to Event-free Survival Event
Description: Event-free survival was defined as the time between randomization and the date of disease progression, relapse, start of new Chronic Lymphocytic Leukemia treatment or death by any cause.
Time Frame: Median observation time was approximately 66.4 months
Population: Participants from the Intent-to-treat population, that included all randomized participants, with disease progression, relapse, start of new Chronic Lymphocytic Leukemia treatment or death.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 301 | 257
Days | 951.0 [843 to 1039] | 1666.0 [1415 to 1799]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p < .0001, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI [0.48 to 0.67]

8. Secondary Outcome: Final Analysis: Time to Disease-free Survival (DFS) Event in Participants With Complete Response (CR)
Description: CR is defined by at least 8 weeks of: 1)Absence of lymphadenopathy 2)No hepatomegaly or splenomegaly 3)Absence of B-symptoms 4)Normal blood count 5)Bone marrow aspirate and biopsy 8 weeks after the clinical and laboratory results demonstrated that a CR was achieved. A marrow sample had to be normocellular for age with less than 30% lymphocytes. Lymphoid nodules had to be absent. If marrow was hypocellular,a repeat biopsy was taken 4 weeks later and samples were re-reviewed in conjunction with the prior pathology. DFS was calculated from time of CR to relapse or death
Time Frame: Median observation time was approximately 66.4 months
Population: Participants from the Intent-to-treat population, all randomized participants, with complete response who experienced a disease free survival event (disease relapse or death).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 58 | 97
Days | 1488.0 [1198 to 1836] | 1854.0 [1646 to 2208]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p = 0.0523, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.52 to 1.02]

9. Secondary Outcome: Final Analysis: Duration of Response
Description: Duration of response was defined as the time from the first documented Complete Response, Partial Response to disease progression or death by any cause.
Time Frame: Median observation time was approximately 66.4 months
Population: Participants from the Intent-to-treat population, all randomized participants, with complete response or partial response who experienced an event (disease progression or death due to any cause).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 214 | 207
Days | 1102.0 [977 to 1249] | 1718.0 [1618 to 1859]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p < .0001, Log Rank; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.48 to 0.71]

10. Secondary Outcome: Final Analysis: Percentage of Participants With Complete Response (CR) and Partial Response
Description: CR is defined by at least 8 weeks of: 1)Absence of lymphadenopathy 2)No hepatomegaly or splenomegaly 3)Absence of B-symptoms 4)Normal blood count 5)Bone marrow aspirate and biopsy 8 weeks after the clinical and laboratory results demonstrated that a CR was achieved. A marrow sample had to be normocellular for age with less than 30% lymphocytes. Lymphoid nodules had to be absent. If marrow was hypocellular,a repeat biopsy was taken 4 weeks later and samples were re-reviewed in conjunction with the prior pathology. Partial response is defined as a decrease in the size of a tumor, or in the extent of cancer in the body, in response to treatment.
Time Frame: Median observation time was approximately 66.4 months
Population: Intent-to-treat population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 409 | 408
Percentage of participants | 72.4 [67.8 to 76.7] | 85.8 [82.0 to 89.0]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p < .0001, Chi-squared; Odds Ratio (OR) = 2.30, 95% CI 2-sided [1.62 to 3.28]

11. Secondary Outcome: Final Analysis: Time to New Treatment for Chronic Lymphocytic Leukemia(CLL)
Description: The time from randomization to the start of a new treatment.
Time Frame: Median observation time was approximately 66.4 months
Population: Participants from the Intent-to-treat population, that included all randomized participants, who started a new CLL treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Number analyzed (Participants) | 251 | 206
Days | 1455.0 [1324 to 1577] | 2082.0 [1926 to 2253]
Statistical Analysis 1: Comparison: Fludarabine+Cyclophosphamide (FC) vs Fludarabine+Cyclophosphamide+Rituximab (FCR); Test type: Superiority or Other; p < .0001, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.49 to 0.72]

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded until 28 days after completion of study treatment (median time approximately 21 months). Serious Adverse Events reported until 1 year post-treatment or initiation of new CLL treatment (median time approximately 42 months).
Description: The safety population included all participants who received at least one dose of study drug.
Arm/Group | Fludarabine+Cyclophosphamide (FC) | Fludarabine+Cyclophosphamide+Rituximab (FCR)
Serious Adverse Events (participants affected / at risk) | 164/398 | 186/402
Other Adverse Events (participants affected / at risk) | 122/398 | 185/402
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine+Cyclophosphamide (FC) (N=398) | Fludarabine+Cyclophosphamide+Rituximab (FCR) (N=402)
Pneumonia (Infections and infestations) | 21 | 18
Herpes Zoster (Infections and infestations) | 6 | 8
Sepsis (Infections and infestations) | 8 | 5
Bronchitis (Infections and infestations) | 5 | 5
Infection (Infections and infestations) | 2 | 5
Gastroenteritis (Infections and infestations) | 3 | 2
Sinusitis (Infections and infestations) | 1 | 4
Erysipelas (Infections and infestations) | 1 | 2
Hepatitis B (Infections and infestations) | 2 | 1
Pneumocystis Jiroveci Infection (Infections and infestations) | 1 | 2
Pneumocystis Jiroveci Pneumonia (Infections and infestations) | 1 | 2
Pneumonia Primary Atypical (Infections and infestations) | 1 | 2
Viral Infection (Infections and infestations) | 0 | 3
Cellulitis (Infections and infestations) | 1 | 1
Cerebral Toxoplasmosis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 2
Neutropenic Infection (Infections and infestations) | 0 | 2
Oral Herpes (Infections and infestations) | 2 | 0
Pneumonia Fungal (Infections and infestations) | 1 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Chronic Sinusitis (Infections and infestations) | 1 | 0
Cytomegalovirus Infection (Infections and infestations) | 0 | 1
Enterococcal Bacteraemia (Infections and infestations) | 0 | 1
Gastroenteritis Cryptosporidial (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Hepatobiliary Infection (Infections and infestations) | 1 | 0
Herpes Simplex (Infections and infestations) | 0 | 1
Herpes Virus Infection (Infections and infestations) | 0 | 1
Herpes Zoster Ophthalmic (Infections and infestations) | 1 | 0
Infected Skin Ulcer (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1
Lung Infection Pseudomonal (Infections and infestations) | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 1 | 0
Oesophageal Candidiasis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 0 | 1
Periorbital Cellulitis (Infections and infestations) | 0 | 1
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 1 | 0
Pseudomonal Sepsis (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 0 | 1
Skin Infection (Infections and infestations) | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 22 | 31
Anaemia (Blood and lymphatic system disorders) | 10 | 6
Leukopenia (Blood and lymphatic system disorders) | 3 | 9
Neutropenia (Blood and lymphatic system disorders) | 3 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 6
Pancytopenia (Blood and lymphatic system disorders) | 3 | 7
Haemolysis (Blood and lymphatic system disorders) | 3 | 1
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 0 | 3
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 2
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 | 1
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 | 0
Coombs Positive Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Evans Syndrome (Blood and lymphatic system disorders) | 1 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Pyrexia (General disorders) | 20 | 18
Chest Pain (General disorders) | 1 | 3
Chills (General disorders) | 0 | 2
Adverse Drug Reaction (General disorders) | 0 | 1
Chest Discomfort (General disorders) | 0 | 1
Death (General disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 1 | 0
General Symptom (General disorders) | 1 | 0
Ill-Defined Disorder (General disorders) | 1 | 0
Mucosal Inflammation (General disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 2 | 1
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung Squamous Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central Nervous System Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Histiocytosis Haematophagic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma Transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pharyngeal Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alveolitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea at Rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiration Abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 2 | 5
Cardiac Failure (Cardiac disorders) | 1 | 1
Coronary Artery Disease (Cardiac disorders) | 2 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 2
Myocardial Ischaemia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 2
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Cardiopulmonary Failure (Cardiac disorders) | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 0 | 1
Supraventricular Extrasystoles (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Ventricular Fibrillation (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 5
Vomiting (Gastrointestinal disorders) | 2 | 3
Abdominal Pain (Gastrointestinal disorders) | 3 | 1
Inguinal Hernia (Gastrointestinal disorders) | 1 | 1
Abdominal Symptom (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Ulcer (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Tongue Ulceration (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 1 | 2
Cerebrovascular Accident (Nervous system disorders) | 0 | 2
Convulsion (Nervous system disorders) | 0 | 1
Diabetic Neuropathy (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Optic Neuritis (Nervous system disorders) | 0 | 1
Stupor (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 1
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 1 | 1
Leukocytoclastic Vasculitis (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pustular Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Hepatic Siderosis (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 3
Drug Hypersensitivity (Immune system disorders) | 0 | 2
Anaphylactic Reaction (Immune system disorders) | 0 | 1
Cytokine Release Syndrome (Immune system disorders) | 0 | 1
Retinal Detachment (Eye disorders) | 1 | 1
Amaurosis Fugax (Eye disorders) | 0 | 1
Dacryostenosis Acquired (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 0 | 1
Vitreous Haemorrhage (Eye disorders) | 1 | 0
Catheterisation Cardiac (Investigations) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Coronary Revascularisation (Surgical and medical procedures) | 1 | 0
Haemorrhoid Operation (Surgical and medical procedures) | 1 | 0
Prostatectomy (Surgical and medical procedures) | 0 | 1
Surgery (Surgical and medical procedures) | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Body Temperature Increased (Investigations) | 0 | 1
Completed Suicide (Psychiatric disorders) | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0
Calculus Ureteric (Renal and urinary disorders) | 1 | 2
Cystitis Haemorrhagic (Renal and urinary disorders) | 0 | 2
Renal Failure (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 2
Deep Vein Thrombosis (Vascular disorders) | 2 | 0
Circulatory Collapse (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Vasculitis Necrotising (Vascular disorders) | 0 | 1
Venous Thrombosis Limb (Vascular disorders) | 0 | 1
Device related infection (Infections and infestations) | 1 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 1
Device occlusion (General disorders) | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Endophthalmitis (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine+Cyclophosphamide (FC) (N=398) | Fludarabine+Cyclophosphamide+Rituximab (FCR) (N=402)
Neutropenia (Blood and lymphatic system disorders) | 71 | 116
Leukopenia (Blood and lymphatic system disorders) | 45 | 88
Thrombocytopenia (Blood and lymphatic system disorders) | 35 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.